CLINICAL TRIAL: NCT03500120
Title: Case Detection and Confirmation, Subtype Classification of Patients With Primary Aldosteronism
Brief Title: Diagnostic Accuracy of Seated Saline Suppression Test for Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, M.D., PhD, Chongqing Medical University
Other Study IDs: DASSSTPA 2017
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2020-04

CONDITIONS: Primary Aldosteronism
Keywords: Saline suppression testing, Seated, Recumbent
MeSH Terms: conditions — Hyperaldosteronism; Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and complete blood cell. Application: 1. diagnosis of PA and primary hypertension; 2.differential diagnosis of PA;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Aldosteronism: Aldosterone/renin concentration ratio(ARR)≥1.0 (ng/dl)/(mIU/l) and 2. PAC post-FST≥6 ng/dl
  Interventions: Diagnostic Test: Seated saline infusion test
- non Primary Aldosteronism: 1. ARR≥1.0 (ng/dl)/(mIU/l) and 2. PAC post-FST<6 ng/dl
  Interventions: Diagnostic Test: Seated saline infusion test

INTERVENTIONS:
Diagnostic Test: Seated saline infusion test — Seated saline infusion test: All participants received the infusion of 2 liters of 0.9% saline over 4 h in seated posture.
  Fludrocortisone suppression test:Patients received 0.1 mg oral fludrocortisone every 6 h for 4 days, together with slow-release potassium chloride and sodium chloride supplements.
  Captopril challenge test:Patients received 50 mg captopril orally at 8-9 a.m. after sitting or standing for at least 1 h. Blood samples were drawn at time zero and 2 h after the challenge.
  Other Names: Captopril challenge test; Fludrocortisone suppression test

SUMMARY:
The present study was undertaken prospectively to compare the diagnostic significance of the seated saline suppression testing (SSST) with the captopril challenge testing (CCT) in hypertensive patients with suspected primary aldosteronism (PA) using the fludrocortisone suppression testing (FST) as the reference standard, and to investigate the optimal cutoff of SSST for differentiating PA from other forms of hypertension.

DETAILED DESCRIPTION:
The diagnosis of primary aldosteronism (PA) typically requires at least one confirmatory test. Four tests are commonly recommended by the Endocrine Society guideline, namely, oral sodium loading, saline infusion, fludrocortisone administration with oral sodium loading, and captopril challenge testing (CCT). Of these, fludrocortisone suppression testing (FST) has been considered the most reliable, but is cumbersome, difficult to perform, and relatively expensive, requiring hospital admission for several days. Alternative approaches to FST have included saline suppression testing (SST), Which requiring patients staying in the recumbent position for at least 1 h before and during the infusion of 2 L of 0.9% saline IV over 4 h. This approach also has the disadvantages of brings much inconvenience to the patient (such as urination or defecation, etc.). Ashraf H. et al. have reported that seated SST (SSST) is more sensitive than recumbent SST (RSST), especially for posture-responsive PA (95.8% versus 33.3%), however, in this small scale study, only 31 patients was PA and only three patients was tested negative for PA by FST. Specificity of each form of SST was unable to estimate and meaningful receiver operating characteristic (ROC) curve analyses could not be performed. Furthermore, it is lack of study in Chinese people. In addition, the investigators have previously found the CCT was as accurate as the FST and plasma aldosterone concentration (PAC) post-CCT is the best approach to interpret the results of the CCT. The present study was undertaken prospectively to compare the diagnostic significance of the SSST with the CCT in hypertensive patients with suspected PA using the FST as the reference standard, and to investigate the optimal cutoff of SSST for differentiating PA from other forms of hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. patients with Joint National Commission stage 2 (>160-179/100-109mm Hg), stage 3 (>180/110 mmHg), or drug-resistant hypertension;
2. hypertension and spontaneous or diuretic-induced hypokalemia;
3. hypertension with adrenal incidentaloma;
4. hypertension and a family history of early-onset hypertension;
5. cerebrovascular accident at a young age (<40 years);
6. all hypertensive first-degree relatives of patients with PA.

Exclusion Criteria:

1. heart failure;
2. chronic kidney disease with an estimated Glomerular Filtration Rate <30 ml/min/1.73 m2;
3. liver cirrhosis;
4. terminal malignant tumor;
5. current use of steroids or oral contraceptives;
6. pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital or clinic patients with hypertension in a single tertiary hospital center.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Seated Saline Suppression Test | 2 weeks
  compare the diagnostic significance of the SSST with the CCT in hypertensive patients with suspected PA using the FST as the reference standard

SECONDARY OUTCOMES:
The cutoff of SSST for diagnosis of PA | 2 weeks
  investigate the optimal cutoff of SSST for differentiating PA from other forms of hypertension.

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, PHD, Study Chair — the Chongqing Primary Aldosteronism Study (CONPASS) Group
Locations (1):
- The First Affilated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nishikawa T, Omura M, Satoh F, Shibata H, Takahashi K, Tamura N, Tanabe A; Task Force Committee on Primary Aldosteronism, The Japan Endocrine Society. Guidelines for the diagnosis and treatment of primary aldosteronism--the Japan Endocrine Society 2009. Endocr J. 2011;58(9):711-21. doi: 10.1507/endocrj.ej11-0133. Epub 2011 Aug 9. PMID 21828936
- [Background] Reznik Y, Amar L, Tabarin A. SFE/SFHTA/AFCE consensus on primary aldosteronism, part 3: Confirmatory testing. Ann Endocrinol (Paris). 2016 Jul;77(3):202-7. doi: 10.1016/j.ando.2016.01.007. Epub 2016 Jun 16. PMID 27318644
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Mulatero P, Dluhy RG, Giacchetti G, Boscaro M, Veglio F, Stewart PM. Diagnosis of primary aldosteronism: from screening to subtype differentiation. Trends Endocrinol Metab. 2005 Apr;16(3):114-9. doi: 10.1016/j.tem.2005.02.007. PMID 15808809
- [Result] Mulatero P, Milan A, Fallo F, Regolisti G, Pizzolo F, Fardella C, Mosso L, Marafetti L, Veglio F, Maccario M. Comparison of confirmatory tests for the diagnosis of primary aldosteronism. J Clin Endocrinol Metab. 2006 Jul;91(7):2618-23. doi: 10.1210/jc.2006-0078. Epub 2006 May 2. PMID 16670162
- [Result] Ahmed AH, Cowley D, Wolley M, Gordon RD, Xu S, Taylor PJ, Stowasser M. Seated saline suppression testing for the diagnosis of primary aldosteronism: a preliminary study. J Clin Endocrinol Metab. 2014 Aug;99(8):2745-53. doi: 10.1210/jc.2014-1153. Epub 2014 Apr 24. PMID 24762111